CLINICAL TRIAL: NCT03555136
Title: Real-life Effectiveness of Vortioxetine in Patients With Major Depressive Disorder: Non-interventional, Multi-national, Prospective Cohort Study to Assess Real-life Effectiveness of Vortioxetine
Brief Title: Real-life Effectiveness of Vortioxetine in Depression
Acronym: RELIEVE
Status: Completed | Type: Observational
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 17354N
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients initiating vortioxetine treatment: Patients with major depressive disorder initiating treatment with vortioxetine
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Treatment with vortioxetine as per local SmPC

SUMMARY:
Worldwide Major Depressive Disorder (MDD) has significant negative personal, societal and economic consequences.

Vortioxetine (Brintellix®) is a new antidepressant authorized since 2013. Despite evidence generated from clinical trials which demonstrate that vortioxetine is an efficacious, well-tolerated antidepressant, there is a need to determine the effectiveness of vortioxetine in real life routine practice.

The study aim is to examine the real-life effectiveness of vortioxetine on functioning, depressive symptom relief, cognition and quality of life.

This is an observational, multi-national, study in patients with MDD initiating treatment with vortioxetine. Information will be collected by the physician, from the patient and their medical record at three time points - baseline, week 12 and week 24 (end of follow-up). This study will be conducted in six countries. In total 2,100 patients are planned for enrolment.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥18 years
* The patient is an outpatient, treated in a GP or psychiatric outpatient practice
* The patient has a diagnosis of major depressive episode according to local diagnostic criteria
* The patient has been prescribed vortioxetine according to the local Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* The patient is unable to read and understand the information sheet and informed consent form or the Patient Reported Outcomes (PRO)
* The patient is concurrently participating in a clinical trial
* The patient has a diagnosis of schizophrenia or other psychotic disorder according to local diagnostic criteria
* The patient has a diagnosis of bipolar disorder according to local diagnostic criteria
* The patient has a substance use disorders other than tobacco use disorder
* The patient has dementia or other neurodegenerative disease significantly impacting cognitive functioning
* The patient has a mood disorder due to a general medical condition or substances
* The patient is pregnant, ≤6 months post-partum or breastfeeding
* The patient is at significant risk of suicide in the investigator's opinion or the patient has attempted suicide within the last six months
* The patient is a member of the study personnel or of their immediate families, or is a subordinate (or immediate family member of a subordinate) to any of the study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from primary, secondary or tertiary care centres
Sampling Method: Probability Sample
Enrollment: 992 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Sheehan Disability Scale (SDS) | Change since baseline at week 12 and 24
  A series of patient self-rated, scales designed to measure the extent to which his or her 1) work or school, 2) social life or leisure activities, and 3) home life or family responsibilities are impaired by his or her symptoms

SECONDARY OUTCOMES:
The Patient Health Questionnaire - nine items (PHQ-9) | Change since baseline at week 12 and 24
  A patient-rated scale designed to assess depression based on the nine DSM-IV criteria for depression
Perceived Deficits Questionnaire - Depression - five items (PDQ-D-5) | Change since baseline at week 12 and 24
  A self-reported rating scale that aims to assess perceived cognitive deficits from the patient's perspective

CONTACTS AND LOCATIONS:
Overall Officials: Email contact H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (106):
- United States (31):
  - Harmonex Neuroscience Research Inc (US0072), Dothan, Alabama
  - Center For Advanced Improvement (US0011), Tucson, Arizona
  - Pharmacology Research Institute (US0045), Newport Beach, California
  - North County Clinical Research (Nccr) (US0071), Oceanside, California
  - Breakthrough Clinical Trials (US0074), San Bernardino, California
  - Viking Clinical Research Center LLC (US0033), Temecula, California
  - Da Vinci Research Institute (US0063), Boca Raton, Florida
  - Sarkis Clinical Trials (US0066), Gainesville, Florida
  - Maxblue Institute (US0038), Hialeah, Florida
  - Office Of Amit Vijapura, Md (US0057), Jacksonville, Florida
  - International Research Associates LLC (US0060), Miami, Florida
  - Millenia Psychiatry and Research, Inc. (US0015), Orlando, Florida
  - Professional Health Care of Pinellas (US0050), St. Petersburg, Florida
  - Northwest Behavioral Research Center (US0007), Marietta, Georgia
  - Pearl Health Clinic (US0001), Ammon, Idaho
  - Southern Illinois Associates LLC (US0079), Glen Carbon, Illinois
  - AMR- Baber Research, Inc. (US0006), Naperville, Illinois
  - University Of Kansas Cancer Center (US0078), Kansas City, Kansas
  - Neuroscientific Insights (US0029), Rockville, Maryland
  - Rochester Center For Behavioral Medicine (US0059), Rochester Hills, Michigan
  - St. Charles Psychiatric Associates - Midwest Research Group (US0039), Saint Charles, Missouri
  - Alivation Research, LLC (US0020), Lincoln, Nebraska
  - Meridian Clinical Research (US0027), Norfolk, Nebraska
  - Finger Lakes Clinical Research (US0005), Rochester, New York
  - Quest Therapeutics Of Avon Lake (US0002), Avon Lake, Ohio
  - Psychiatric Consultants, Pc (US0028), Franklin, Tennessee
  - Bay Pointe Behavioral Health (US0030), Friendswood, Texas
  - Biopharma Informatic, LLC (US0031), Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - West park Springs (US0073), Richmond, Texas
  - Core Clinical Research (US0067), Everett, Washington
- Canada (10):
  - Chokka Center For Integrative Health (CA0001), Edmonton, Alberta
  - Chatham-Kent Clinical Trials Research Centre (CA0007), Chatham, Ontario
  - Queen's University-Hotel Dieu Hospital (CA0011), Kingston, Ontario
  - St. Joseph's Health Care London - Parkwood Institute (Regional Mental Health Care London and Parkwood Hospital) (CA0004), London, Ontario
  - Start Clinic For Mood And Anxiety Disorders (CA0006), Toronto, Ontario
  - Jodha Tishon Inc (CA0008), Toronto, Ontario
  - GCP Research (CA0013), Montreal, Quebec
  - Mana Research Inc (CA0012), Point Claire, Quebec
  - Alpha Recherche Clinique (CA0009), Québec, Quebec
  - Alpha Recherche Clinique (CA0017), Québec
- France (37):
  - Centre Hospitalier Bp29 (FR0015), Rouffach, Alsace
  - Dr Philippe Marmor, MD, Office of (FR0035), Strasbourg, Alsace
  - CHU de Nantes (FR0023), Nantes, Cedex 1
  - CHS Le Vinatier (FR0013), Bron, Cedex
  - Cmpi (FR0004), Le Vésinet, Yvelines
  - Dr. Philippe Remaud MD, Office of (FR0010), Angers
  - Chru Houtel Dieu (FR0020), Angers
  - Clinique Villa Bleue (FR0008), Angoulême
  - Clinique Clinea orgemont (FR0061), Argenteuil
  - Centre Hospitalier De Blois (FR0011), Blois
  - CH De Novillars (FR0025), Chalezeule
  - CHU Clermont-Ferrand, Hopital Gabriel Montpied (FR0037), Clermont-Ferrand
  - Chs Philippe Pinel (Fr0017), Dury
  - Centre Medical Ambroise Pare (FR0005), Élancourt
  - Hopital Albert Michallon- CHU Grenoble Alpes (FR0021), Grenoble
  - Clinique Korian La Crau (FR0063), La Crau
  - Dr. Norbert Rigaud Md, Office Of (FR0028), Lamagistère
  - Centre Hospitalier Esquirol (FR0038), Limoges
  - Clinique Mon Repos (FR0057), Marseille
  - Centre Hospitalier De Martigues (FR0064), Martigues
  - Hopital de la Colombiere (FR0026), Montpellier
  - Cabinet Medical (FR0043), Mulhouse
  - Maison Des Addictions (FR0006), Nancy
  - Centre Hospitalier Universitaire (CHU) de Nice - Hopital Pasteur - Clinique de Psychiatrie et de Psychologie Medicale (FR0041), Nice
  - Centre Hospitalier Universitaire de Nimes (FR0018), Nîmes
  - Centre Hospitalier Sainte Anne (FR0029), Paris
  - Camp Antonin Artaud (FR0001), Quimper
  - Dr. Dominique Januel, MD Office of (FR0044), Rueil-Malmaison
  - Unites De Soins Romain Rolland (FR0012), Saint-Denis
  - Hopital Nord (FR0042), Saint-Priest-en-Jarez
  - Dr Lousqui Charles MD, Office of (FR0033), Strasbourg
  - Hopital civil (FR0039), Strasbourg
  - Cabinet Du Dr D Bonneau (FR0036), Thouars
  - Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer - Hôpital Sainte Musse (FR0019), Toulon
  - Hopital De Psychiatrie (FR0009), Toulouse
  - Dr. David Modavi Md, Office Of (FR0034), Toulouse
  - Dr. Joel Pon MD, Office of (FR0027), Toulouse
- Italy (28):
  - Ospedale Versilia (IT0002), Lucca, LU
  - Casa di Cura Villa San Benedetto Menni, Suore Ospedaliere (IT0025), Albese Con Cassano, Milano
  - Asl Roma G (IT0005), Colleferro, Roma
  - Ospedale Sant'Andrea Hospital (IT0003), Rome, Roma
  - Insituto Di Ricovero E Cura A Carattere Scientifico San Raffaele Pisana (IT0035), Roma, Rome
  - DSM Giulianova - ospedale di Giulianova (IT0019), Giulianova, Teramo
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga (IT0004), Orbassano, Torino
  - Istituto di Neuroscienze (INS) (IT0028), Florence, Tuscany
  - Azienda Ospedaliera di Perugia - Policlinico Monteluce (IT0034), Perugia, Umbria
  - ASST Papa Giovanni XXIII (IT0016), Bergamo
  - Università degli Studi di Brescia (IT0029), Brescia
  - Universita Degli Studi Di Catania - Azienda Policlinico (IT0030), Catania
  - Universita Degli Studi Magna Graecia Di Catanzaro (IT0006), Catanzaro
  - DSM Cosenza (IT0015), Cosenza
  - Psichiatria Ospedale Oglio Po (IT0023), Cremona
  - Ospedali Riuniti Foggia (IT0007), Foggia
  - Dipartimento Salute Mentale ASL Lecce (IT0009), Lecce
  - ASST Lodi (IT0042), Lodi
  - Azienda Toscana nord ovest zona Apuane (IT0039), Massa
  - Policlinico Universitario Di Messina (IT0031), Messina
  - Azienda Ospedaliera San Paolo - Universita Degli Studi Di Milano (IT0014), Milan
  - Disturbi Depressivi Ospedale Luigi Sacco Polo Universitario Psichiatria 2 - CTDD (IT0033), Milan
  - Pneumology Clinic - AO San Gerardo (IT0017), Monza
  - Universita degli Studi di Roma La Sapienza - Umberto I Policlinico di Roma (IT0032), Roma
  - Villa Von Siebenthal (IT0008), Roma
  - Universita Cattolica del Sacro Cuore (University of Sacred Heart Policlinico A. Gemelli) (IT0018), Rome
  - Ospedale Alfredo Fiorini (IT0026), Terracina
  - University Of Turin (IT0001), Turin

REFERENCES:
- [Derived] Di Nicola M, Adair M, Rieckmann A, Christensen M C. Effectiveness of vortioxetine in elderly patients with major depressive disorder in real-world clinical practice: Results from the RELIEVE study. J Psychopharmacol. 2024 Jul;38(7):615-623. doi: 10.1177/02698811241260996. PMID 39077889
- [Derived] Almeida SS, Christensen MC, Simonsen K, Adair M. Effectiveness of vortioxetine in patients with major depressive disorder and co-morbid generalized anxiety disorder in routine clinical practice: A subgroup analysis of the RELIEVE study. J Psychopharmacol. 2023 Mar;37(3):279-288. doi: 10.1177/02698811221132468. Epub 2022 Nov 15. PMID 36377523